CLINICAL TRIAL: NCT01305239
Title: A Survey Of Clinical Practice Of Adjuvant Treatment Of Breast Cancer Using Exemestane (Aromasin®) In Postmenopausal Hr+ Patients
Acronym: ETAPE
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NRA5990024; A5991095, ETAPE
Record Dates: First submitted 2011-02-24; First posted 2011-02-28 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: Observational; epidemiological; cohort; cross-sectional; prospective; multicenter; survey; France.
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postmenopausal ER+ patients treated by Aromasin.
  Interventions: Drug: Aromasin

INTERVENTIONS:
Drug: Aromasin — Aromasin 25 mg daily.
  Other Names: Exemestane

SUMMARY:
Observational survey aiming to evaluate the tolerability of Aromasin and the ways in which it is used in clinical practice in France (as adjuvant endocrine therapy).

DETAILED DESCRIPTION:
It was hypothesized that 200 participating doctors would provide the survey with sufficient statistical precision to meet the objectives, with each participating doctor recruiting up to 6 patients. An initial sample of 1000 doctors should be contacted (letter, phone).

These 1000 doctors will initially be chosen at random from a file held by Pfizer of doctors who have agreed to take part in a Pfizer survey.

These doctors will be experienced and qualified in the treatment and management of patients with non-metastatic, surgically-treated breast cancer (medical oncologists, gynaecologists, and medical oncologists/ radiation oncologists). They are practicing in general hospitals, teaching hospitals, CRLCC cancer centres and private clinics treating patients with breast cancer.

Study recruitment was stopped due to difficulty in enrolling the targeted number of patients on December 3, 2010. There were no safety concerns involved in the decision to stop enrollment.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal patients, defined as: natural menopause for at least 1 year, surgical ovariectomy, chemotherapy-induced amenorrhoea for at least 2 years.

Patients who have had surgical treatment for histologically confirmed breast cancer that was nonmetastatic at the time of the initial diagnosis.

Patients whose tumour was hormone receptor positive (HR+, ER+ and/or PR+). Patients initiated on Aromasin at least 2 months before inclusion but not more than 1 year.

Exclusion Criteria:

Patients for whom Aromasin treatment is contraindicated. Presence of metastasis or a contralateral tumour. Another adjuvant endocrine therapy. Another concomitant antineoplastic treatment (except for Herceptin®). Participation in a clinical trial with an investigational drug during the 30 days prior to enrolment in the study.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal patients, hormone receptor positive, who have had surgical treatment for histologically confirmed early breast cancer that was nonmetastatic at the time of the initial diagnosis, treated by Aromasin as adjuvant endocrine therapy.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NRA5990024&StudyName=A%20Survey%20Of%20Clinical%20Practice%20Of%20Adjuvant%20Treatment%20Of%20Breast%20Cancer%20Using%20Exemestane%20%28Aromasin%AE%29%20In%20Postmenopausal%20Hr+%20Patients%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: 25 mg oral tablet once a day
Period: Overall Study
Arm/Group | Exemestane
Started | 398
Safety Set | 397
Intent to Treat Population | 287
Completed | 375
Not Completed | 23
Not completed — Adverse Event | 22
Not completed — Exemestane taken prior to inclusion only | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane
Number analyzed (Participants) | 397
Age Continuous [Mean (Standard Deviation); unit: years] — N = 392, number of participants with baseline age data.
  years | 63.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 397
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a patient who received study drug was considered an adverse event without regard to possibility of causal relationship. An adverse event resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a serious adverse event: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline, every 6 months until adjuvant hormonal therapy stopped or up to 5 years of therapy completed
Population: Safety set: all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Exemestane
Number analyzed (Participants) | 397
percentage of participants
  AE | 41.6
  SAE | 0.5

2. Secondary Outcome: Reasons for Discontinuation of Aromasin Therapy
Time Frame: Baseline, every 6 months until adjuvant hormonal therapy stopped or up to 5 years of therapy completed
Population: Safety set. N = number of participants with follow-up visit(s) who discontinued treatment with exemestane.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 45
participants
  Therapeutic choice | 9
  Adverse events | 36

3. Secondary Outcome: Percentage of Participants Who Were Compliant With Treatment
Description: Compliant with treatment = followed treatment regimen with exemestane according to initial prescription.
Time Frame: Baseline, every 6 months until adjuvant hormonal therapy stopped or up to 5 years of therapy completed
Population: Safety set. Information on compliance was not available for subjects who did not have a follow-up visit. N = number of participants with analyzable data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane
Number analyzed (Participants) | 286
percentage of participants | 90.2 [85.3 to 95.1]

4. Secondary Outcome: Duration of Treatment
Description: Total duration of adjuvant hormonal therapy with exemestane.
Time Frame: Baseline, every 6 months until adjuvant hormonal therapy stopped or up to 5 years of therapy completed
Population: Safety set; N = number of participants with analyzable (non-missing) data. For 2 participants lost to follow-up, the duration of exemestane was calculated until the date of lost to follow-up.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Exemestane
Number analyzed (Participants) | 252
months | 15.9 (7.8)

5. Secondary Outcome: Event-free Survival
Description: Event-free survival: time between first intake of exemestane and date of last follow-up or date of death for deceased participants (date of relapse or death or last follow-up minus first intake date) + 1 / 365.25 * 12.
Time Frame: Baseline, every 6 months until adjuvant hormonal therapy stopped or up to 5 years of therapy completed
Population: ITT population = all participants who received at least 1 dose of study drug and had at least 1 follow-up questionnaire completed. N = number of participants with analyzable (non-missing) data.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Exemestane
Number analyzed (Participants) | 251
months | 16.2 [13.9 to 18.4]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 2/397
Other Adverse Events (participants affected / at risk) | 173/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=397)
Cardiac failure (Cardiac disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=397)
Arrhythmia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oral discomfort (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 2
Chest discomfort (General disorders) | 1
Fatigue (General disorders) | 51
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Sense of oppression (General disorders) | 1
Cystitis escherichia (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 3
Scapula fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2
Quality of life decreased (Investigations) | 2
Weight increased (Investigations) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic disorder (Metabolism and nutrition disorders) | 3
Missing code (General disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 89
Back pain (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 34
Osteoporosis (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 17
Insomnia (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 4
Libido disorder (Psychiatric disorders) | 14
Sexual inhibition (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Breast discomfort (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 1
Genital disorder female (Reproductive system and breast disorders) | 4
Menometrorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dialysis (Surgical and medical procedures) | 1
Axillary vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 59
Hypertension (Vascular disorders) | 7
Phlebitis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Study recruitment was stopped due to difficulty enrolling the target number of participants. There were no safety concerns in the decision to terminate this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.